CLINICAL TRIAL: NCT00642551
Title: Clinical Trial on Beneficial Effects of Long Term Menaquinone-7 (Vitamin K2) Intake by Postmenopausal Women
Brief Title: Beneficial Effects of Long Term Menaquinone-7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 07-3-074
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Bone Loss; Arteriosclerosis
Keywords: vitamin K2; menaquinone-7; bone health; vascular health
MeSH Terms: conditions — Bone Diseases, Metabolic; Arteriosclerosis | interventions — menaquinone 7

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-7 (Active Comparator): 1 capsule per day existing of 180 µg menaquinone-7
  Interventions: Dietary Supplement: menaquinone-7
- Placebo (Placebo Comparator): 1 placebo capsule per day for three years
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: menaquinone-7 — 180 µg menaquinone-7 daily for three years
  Arms: MK-7
Dietary Supplement: placebo — 1 placebo capsule daily for three years
  Arms: Placebo

SUMMARY:
From all K-vitamins, menaquinone-7 (MK-7) has been identified now as the most effective cofactor for the carboxylation reaction of Gla-proteins such as osteocalcin (in bone) and matrix-Gla protein (in the arterial vessel wall). The question remains whether supplementation with MK-7 also leads to measurable improvements of bone and vascular health. The purpose of the study is to demonstrate that MK-7 has a health benefit in apparently healthy postmenopausal women. In a placebo-controlled randomized clinical trial the effect of an MK-7- supplement will be monitored during three years on bone quantity and quality and on vascular characteristics and function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women between 55 and 65 years old
* Subjects of normal body weight and height according to BMI < 30
* Subjects of Caucasian race
* Subject has given written consent to take part in the study

Exclusion Criteria:

* Subjects with (a history of) metabolic or gastrointestinal disease
* Subjects presenting chronic degenerative and/or inflammatory disease
* Subjects receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters
* Subjects receiving corticoϊd treatment
* Subjects using oral anticoagulants
* Subject using bisphosphonates
* Subjects using hormone replacement therapy
* Subjects undergoing ovariectomy and/or hysterectomy
* Subject with (a history of) soy allergy
* Subjects using vitamin K containing multivitamins or vitamin K supplements
* Subjects who have participated in a clinical study more recently than one month before the current study
* Subjects who are found to be osteoporotic at baseline (T-score < -2.5)

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Bone mineral density, bone mineral content and bone geometry measured by DEXA. Vascular elasticity, intima-media thickness and pulse wave velocity measured by ultrasound | three years

SECONDARY OUTCOMES:
The vitamin K-dependent proteins: uncarboxylated osteocalcin (ucOC), carboxylated osteocalcin (cOC), uncarboxylated matrix-Gla protein (ucMGP) and carboxylated matrix-Gla protein cMGP) | three years

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — Maastricht University
Locations (1):
- VitaK BV / Maastricht University, Maastricht, PO Box 616, Netherlands

REFERENCES:
- [Derived] Knapen MH, Schurgers LJ, Shearer MJ, Newman P, Theuwissen E, Vermeer C. Association of vitamin K status with adiponectin and body composition in healthy subjects: uncarboxylated osteocalcin is not associated with fat mass and body weight. Br J Nutr. 2012 Sep 28;108(6):1017-24. doi: 10.1017/S000711451100626X. Epub 2011 Dec 5. PMID 22136751